CLINICAL TRIAL: NCT00596752
Title: Multinational, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel Groups Study to Assess the Efficacy and Safety of Prostaglandin E1 in Subjects With Critical Limb Ischemia (Fontaine Stage IV)
Brief Title: Alprostadil in Peripheral Arterial Occlusive Disease (PAOD) Stage IV
Acronym: ESPECIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Aptiv Solutions (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0777; 2005-001970-29 (EudraCT Number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-17 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Alprostadil; Prostavasin; PAOD; Fontaine Stage IV
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Alprostadil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alprostadil (Experimental): Prostavasin® 40 μg will be infused intravenously twice daily over 2 hours in 50 to 150 ml isotonic sodium chloride solution during a Treatment Phase of 4 weeks.
  Interventions: Drug: Alprostadil
- Placebo (Placebo Comparator): Placebo will be infused intravenously twice daily over 2 hours in 50 to 150 ml isotonic sodium chloride solution during a Treatment Phase of 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alprostadil — * Active Substance: Prostaglandin E1
  * Pharmaceutical Form: solution for infusion
  * Concentration: 40 μg b.d.
  * Route of Administration: intravenous infusion
  Other Names: Prostavasin
  Arms: Alprostadil
Other: Placebo — * Active Substance: Lactose
  * Pharmaceutical Form: solution for infusion
  * Concentration: 40 μg b.d.
  * Route of Administration: intravenous infusion
  Arms: Placebo

SUMMARY:
The study is to confirmatorily show a superior effect of Alprostadil compared to placebo on the rate of complete healing of ischemic necroses and ulcerations as well as on the frequency and height of major amputations in patients suffering from PAOD stage IV.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 45 years of age
* Subjects with macro-angiopathy, proven PAOD Stage IV with up to 2 ischaemic skin lesions for more than 2 weeks
* Subject has a complete angiography of pelvis, thigh and calf within one month of inclusion
* Systolic ankle pressure ≤ 70 mmHg in subjects without media sclerosis of the lower limb artery or systolic big toe pressure ≤ 50 mmHg in diabetics with media sclerosis of the lower limb artery
* Subject is not in the position to be primarily revascularized or refuses surgery

Exclusion Criteria:

* Imminent or foreseeable amputation
* Major amputation on the affected extremity
* History of chronic alcohol or drug abuse
* More than two ischemic ulcerations
* One ulcer ≥ 6 cm^2, both ulcers ≤ 1 cm^2 or at least one ulcer affecting the bone or tendons
* Acute ischemia and peripheral vascular disorders of inflammatory or immunologic origin
* Neuropathic or venous ulcers
* Buerger's disease
* Septic gangrene
* Use of vasoactive medication or prostaglandins
* Treatment with prostanoids within 3 months prior to inclusion
* Surgical or interventional measures performed on the affected extremity within 3 months prior to study drug treatment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2004-03; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (78):
- Czechia (2):
  - 404, Pilsen
  - 414, Ústí nad Labem
- 1, Karlsbad, Germany
- Mexico (3):
  - 502, Aguascalientes
  - 505, Mérida
  - 501, Querétaro
- Poland (16):
  - 306, Bydgoszcz
  - 321, Gmina Końskie
  - 320, Krakow
  - 314, Lublin
  - 315, Lublin
  - 316, Poznan
  - 317, Poznan
  - 301, Szczecin
  - 304, Szczecin
  - 307, Warsaw
  - 308, Warsaw
  - 309, Warsaw
  - 318, Warsaw
  - 319, Warsaw
  - 312, Wroclaw
  - 322, Zamość
- Russia (39):
  - 246, Barnaul
  - 205, Chelyabinsk
  - 244, Chelyabinsk
  - 228, Irkutsk
  - 242, Kazan'
  - 227, Kemerovo
  - 201, Moscow
  - 202, Moscow
  - 203, Moscow
  - 209, Moscow
  - 219, Moscow
  - 220, Moscow
  - 230, Moscow
  - 248, Moscow
  - 231, Novosibirsk
  - 232, Novosibirsk
  - 222, Omsk
  - 217, Petrozavodsk
  - 206, Rostov-on-Don
  - 225, Rostov-on-Don
  - 236, Rostov-on-Don
  - 239, Rostov-on-Don
  - 224, Ryazan
  - 210, Saint Petersburg
  - 212, Saint Petersburg
  - 213, Saint Petersburg
  - 214, Saint Petersburg
  - 215, Saint Petersburg
  - 216, Saint Petersburg
  - 218, Samara
  - 237, Saratov
  - 243, Tula
  - 234, Tver'
  - 238, Tyumen
  - 241, Ufa
  - 240, Volgograd
  - 221, Yaroslavl
  - 223, Yekaterinburg
  - 247, Yekaterinburg
- Ukraine (17):
  - 112, Dnipropetrovsk
  - 109, Donetsk
  - 110, Donetsk
  - 114, Ivano-Frankivsk
  - 111, Kharkiv
  - 101, Kiev
  - 102, Kiev
  - 103, Kiev
  - 104, Kiev
  - 105, Kiev
  - 106, Lviv
  - 118, Odesa
  - 119, Odesa
  - 113, Uzhhorod
  - 116, Vinnytsia
  - 107, Zaporizhzhya
  - 108, Zaporizhzhya

REFERENCES:
- [Result] Lawall H, Pokrovsky A, Checinski P, Ratushnyuk A, Hamm G, Randerath O, Grieger F, Bentz JWG. Efficacy and Safety of Alprostadil in Patients with Peripheral Arterial Occlusive Disease Fontaine Stage IV: Results of a Placebo Controlled Randomised Multicentre Trial (ESPECIAL). Eur J Vasc Endovasc Surg. 2017 Apr;53(4):559-566. doi: 10.1016/j.ejvs.2016.12.035. Epub 2017 Feb 8. PMID 28189475
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in March 2004 in order to end up with 840 enrolled subjects. The study was conducted using a two-stage group sequential adaptive design with possible sample size adjustment after the planned interim analysis, which was performed after stage 1. After the interim analysis subjects were included in stage 2.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS). RS consists of all subjects randomized into the study who have completed the study or terminated prematurely.
Groups:
- Alprostadil: Prostavasin® 40 μg will be infused intravenously twice daily over 2 hours in 50 to 150 ml isotonic sodium chloride solution during a Treatment Phase of 4 weeks.
  Alprostadil: - Active Substance: Prostaglandin E1
  * Pharmaceutical Form: solution for infusion
  * Concentration: 40 μg b.d.
  * Route of Administration: intravenous infusion
- Placebo: Placebo will be infused intravenously twice daily over 2 hours in 50 to 150 ml isotonic sodium chloride solution during a Treatment Phase of 4 weeks.
  Placebo: - Active Substance: Lactose
  * Pharmaceutical Form: solution for infusion
  * Concentration: 40 μg b.d.
  * Route of Administration: intravenous infusion
Period: Overall Study
Arm/Group | Alprostadil | Placebo
Started | 415 | 425
Randomized and Treated | 415 | 424
Completed | 289 | 282
Not Completed | 126 | 143
Not completed — Other Reason | 44 | 49
Not completed — Adverse Event | 34 | 34
Not completed — Lost to Follow-up | 22 | 38
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Unsatisfactory Compliance | 9 | 6
Not completed — Lack of Efficacy | 4 | 7
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set including all randomized subjects who received at least one dose of trial medication. Subjects were analyzed according to the actual treatment received. 4 PBO subjects were treated with Alprostadil, 3 Alprostadil subjects were treated with PBO.1 PBO subject withdrew prior to start of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alprostadil | Placebo | Total
Number analyzed (Participants) | 416 | 423 | 839
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 153 | 170 | 323
  >=65 years | 263 | 253 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.5) | 66.4 (9.3) | 66.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 117 | 240
  Male | 293 | 306 | 599
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 75.4 (11.9) | 76.6 (12.6) | 76.0 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Complete Healing of Ischemic Necroses and Ulcerations at 12 Weeks After the End of Study Drug Treatment
Description: The assessment of ulcer area was collected per lesion with up to 2 lesions per subject (both legs could be affected). In the analysis a subject is only considered completely healed at a time point, if all ischemic lesions are reported as completely healed at that time point.
Time Frame: At 12 weeks after the end of study drug treatment
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF) in case of missing values. FAS consists of all randomized subjects who received at least one dose of trial medication and who provide valid data to assess at least one of the primary efficacy endpoints.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 414 | 424
participants
  Stage 1 (n=253, n=251) | 49 | 43
  Stage 2 (n=161, n=173) | 27 | 30
Statistical Analysis 1: Comparison: Alprostadil vs Placebo; Primary goal was to test the following null hypothesis: H01: πhealingPGE1≤ πhealingPlacebo, with πhealing=proportion of subjects with complete ulcer healing. The planned information rate for stage 1 of the two-stage group sequential test design with an overall one-sided comparison-wise α=0.0125 for this co-primary endpoint is given by 0.83. This is the statistical analysis of stage 1; Test type: Superiority or Other; p = 0.2587, Cochran-Mantel-Haenszel — For confirmatory hypothesis testing the p-values of the normal approximation test for comparing two rates was used as input for the weighted inverse normal method. The 1-sided boundary p-value for stage 1 is given by p1=0.00587; The 2 primary endpoints were tested at one-sided 0.0125 each so that the overall type I error rate of 0.025 was controlled in a strong sense
Statistical Analysis 2: Comparison: Alprostadil vs Placebo; Primary goal was to test the following null hypothesis: H01: πhealingPGE1≤ πhealingPlacebo, with πhealing=proportion of subjects with complete ulcer healing. This is the statistical analysis of stage 1 and stage 2 combined; Test type: Superiority or Other; p = 0.3463, Cochran-Mantel-Haenszel — For confirmatory hypothesis testing the p-values of the normal approximation test for comparing two rates was used as input for the weighted inverse normal method. The 1-sided boundary p-value for stage 1 and 2 combined is given by p2=0.01085; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Occurrence of Major Amputations at 24 Weeks After the End of Study Drug Treatment
Description: Assessment of amputations was collected per leg affected by a lesion with up to 2 lesions per subject. Amputations were regarded as major if they were performed at the ankle joint level or above. Amputations of toes or part of the foot leaving a stump thereon the subject can walk were regarded as minor. An affected leg is defined as a leg with at least 1 lesion on Study Day -6 to -2 and only amputations of affected legs are considered in the efficacy analysis of amputations. A subject is counted as major/minor amputated, if at least 1 affected leg was major/minor amputated.
Time Frame: At 24 weeks after the end of study drug treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 414 | 424
participants
  Stage 1 (n=253, n=251) | 32 | 49
  Stage 2 (n=161, n=173) | 20 | 13
Statistical Analysis 1: Comparison: Alprostadil vs Placebo; Primary goal was to test the following null hypothesis: H02: πampPGE1≥ πampPlacebo, with πamp=proportion of subjects with major amputations. The planned information rate for stage 1 of the two-stage group sequential test design with an overall one-sided comparison-wise α=0.0125 for this co-primary endpoint is given by 0.83. This is the statistical analysis of stage 1; Test type: Superiority or Other; p = 0.0173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alprostadil vs Placebo; Primary goal was to test the following null hypothesis: H02: πampPGE1≥ πampPlacebo, with πamp=proportion of subjects with major amputations. This is the statistical analysis of stage 1 and stage 2 combined; Test type: Superiority or Other; p = 0.1154, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Complete Healing of Ischemic Necroses and Ulcerations at 24 Weeks After the End of Study Drug Treatment
Description: as for outcome 1
Time Frame: At 24 weeks after the end of study drug treatment
Population: Of the 838 subjects in the Full Analysis Set (FAS), 568 are included in the analysis of this outcome measure. FAS consists of all randomized subjects who received at least one dose of trial medication and who provide valid data to assess at least one of the primary efficacy endpoints.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 289 | 279
participants | 108 | 103

4. Secondary Outcome: Intensity of Rest Pain Induced by Ischemic Lesions at 24 Weeks After the End of Study Drug Treatment
Description: Visit values of intensity of rest pain from a visual analogue scale, ranging from 0 mm (no pain) to 100 mm (maximum conceivable pain), had to be reported in the case of presence of rest pain only. If the leading question in regard to the presence of rest pain is answered with "No" and no visit value is specified, the visit value will be set to 0 for the analysis.
Time Frame: At 24 weeks after the end of study drug treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 414 | 424
millimeters (mm) | 17.57 (25.33) | 16.38 (25.08)

5. Secondary Outcome: Increase/Decrease in Ulcer Area of ≥ 50 % at 24 Weeks After the End of Study Drug Treatment
Description: In case of two ulcers the worse ulcer status is analyzed. The categories of investigator assessment are: complete healing, decrease by ≥ 50 %, unchanged, increase by ≥ 50 %.
Time Frame: At 24 weeks after the end of study drug treatment
Population: Of the 838 subjects in the Full Analysis Set (FAS), 465 are included in the analysis of this outcome measure. FAS consists of all randomized subjects who received at least one dose of trial medication and who provide valid data to assess at least one of the primary efficacy endpoints.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 233 | 232
participants
  Complete healing | 101 | 98
  Decrease by >= 50 % | 57 | 56
  Remains unchanged | 45 | 48
  Increase by >= 50 % | 30 | 30

6. Secondary Outcome: Consumption and Type of Analgesic Medication During the Course of the Study (up to 196 Days)
Description: The number of subjects who used analgesics are summarized for different time points/intervals during the course of the study.
Time Frame: During the course of the study (up to 196 days)
Population: Full Analysis Set (FAS) consists of all randomized subjects who received at least one dose of trial medication and who provide valid data to assess at least one of the primary efficacy endpoints.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 414 | 424
participants
  Prior to treatment (n=414, n=424) | 300 | 318
  Concomitant, Study Day 1 (n=414, n=424) | 292 | 314
  Concomitant, Study Day 2 (n=414, n=424) | 295 | 313
  Concomitant, Study Day 3 (n=413, n=424) | 295 | 317
  Concomitant, Study Day 4 (n=412, n=423) | 292 | 316
  Concomitant, Study Day 5 (n=411, n=423) | 294 | 311
  Concomitant, Study Day 6 (n=411, n=423) | 290 | 312
  Concomitant, Study Day 7 (n=409, n=422) | 290 | 306
  Concomitant, Week 2 (n=409, n=422) | 292 | 308
  Concomitant, Week 3 (n=399, n=416) | 259 | 284
  Concomitant, Week 4 (n=393, n=404) | 238 | 257
  Post treatment, Study Days 29-42 (n=348, n=354) | 170 | 191
  Post treatment, Study Days 43-56 (n=361, n=370) | 164 | 173
  Post treatment, Study Days 57-70 (n=361, n=346) | 155 | 155
  Post treatment, Study Days 71-84 (n=352, n=344) | 146 | 148
  Post treatment, Study Days 85-98 (n=341, n=339) | 143 | 140
  Post treatment, Study Days 99-112 (n=321, n=318) | 132 | 127
  Post treatment, Study Days 113-140 (n=309, n=301) | 122 | 117
  Post treatment, Study Days 141-168 (n=306, n=304) | 118 | 109
  Post treatment, Study Days 169-196 (n=272, n=271) | 98 | 90

7. Secondary Outcome: Systolic Pressure at Ankle Level at 24 Weeks After the End of Study Drug Treatment
Description: Systolic pressure at ankle level was measured at the Arteria tibialis posterior and the Arteria dorsalis pedis. Two individual series of measurements of arterial pressures per subject across the assessed visits were selected for the analysis. For the first analysis (worst change analysis) the series of measurements in the one artery which has the worst change from Baseline at the final measurement was used. For the second analysis (worst value analysis) the series of measurements which has the worst final post-Baseline measurement was used. The series relevant for the analyses was selected from the series for the affected leg or legs only. The selection is 1 out of up to 4 series available per subject. Series without Baseline value and series with at least 1 measurement of more than 150 mmHg were excluded from the selection process due to the suspicion of media sclerosis of the lower limb artery.
Time Frame: At 24 weeks after the end of study drug treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 383 | 394
mmHg
  Worst change analysis | 42.83 (30.16) | 39.47 (28.32)
  Worst value analysis | 39.39 (29.92) | 36.45 (27.19)

8. Secondary Outcome: Minor Amputations at 24 Weeks After the End of Study Drug Treatment
Description: Assessment of amputations was collected per leg affected by a lesion with up to 2 lesions per subject. Amputations were regarded as major if they were performed at the ankle joint level or above. Amputations of toes or part of the foot leaving a stump thereon the subject can walk were regarded as minor. An affected leg is defined as a leg with at least 1 lesion on Study Day -6 to -2 and only amputations of affected legs are considered in the efficacy analysis of amputations. A subject is counted as major/minor amputated, if at least 1 affected leg was major/minor amputated.
  The number of subjects with minor amputation prior to or at 24 weeks after the end of study drug treatment is presented below.
Time Frame: At 24 weeks after the end of study drug treatment
Population: Of the 838 subjects in the Full Analysis Set (FAS), 613 are included in the analysis of this outcome measure. FAS consists of all randomized subjects who received at least one dose of trial medication and who provide valid data to assess at least one of the primary efficacy endpoints.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 316 | 297
participants | 65 | 40

9. Secondary Outcome: Revascularization Procedures at 24 Weeks After the End of Study Drug Treatment
Description: The number of subjects with revascularization prior to or at 24 weeks after the end of study drug treatment is presented below.
Time Frame: At 24 weeks after the end of study drug treatment
Population: Of the 838 subjects in the Full Analysis Set (FAS), 577 are included in the analysis of this outcome measure. FAS consists of all randomized subjects who received at least one dose of trial medication and who provide valid data to assess at least one of the primary efficacy endpoints.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 294 | 283
participants | 6 | 7

10. Secondary Outcome: All-cause Mortality During the Course of the Study (up to 196 Days)
Time Frame: During the course of the study (up to 196 days)
Population: Safety Set consists of all randomized subjects who received at least one dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 416 | 423
participants | 20 | 15

11. Secondary Outcome: Cardiovascular Mortality During the Course of the Study (up to 196 Days)
Time Frame: During the course of the study (up to 196 days)
Population: Safety Set consists of all randomized subjects who received at least one dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 416 | 423
participants | 11 | 14

12. Secondary Outcome: Cardiovascular Morbidity During the Course of the Study (up to 196 Days)
Description: Cardiovascular morbidity is presented as number of subjects with myocardial infarction and/or stroke during the course of the study.
Time Frame: During the course of the study (up to 196 days)
Population: Safety Set consists of all randomized subjects who received at least one dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 416 | 423
participants
  Myocardial infarctions | 5 | 6
  Strokes | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the course of the study from Study Day 0 up to Study Day 196.
Description: Adverse Events refer to the Safety Set. Safety Set consists of all subjects who have completed the study or terminated prematurely and who have received at least 1 dose of study medication.
Arm/Group | Alprostadil | Placebo
Serious Adverse Events (participants affected / at risk) | 87/416 | 62/423
Other Adverse Events (participants affected / at risk) | 61/416 | 62/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprostadil (N=416) | Placebo (N=423)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (3) | 3 (3)
CARDIAC FAILURE (Cardiac disorders) | 3 (3) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 2 (2) | 4 (4)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 3 (3)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 2 (2)
ACUTE RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (2)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 (0) | 1 (1)
NODAL ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)
MESENTERIC ARTERY EMBOLISM (Gastrointestinal disorders) | 0 (0) | 1 (1)
ISCHAEMIC ULCER (General disorders) | 2 (2) | 0 (0)
NECROSIS (General disorders) | 2 (2) | 0 (0)
SUDDEN DEATH (General disorders) | 2 (2) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 3 (3)
PYREXIA (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
WOUND NECROSIS (General disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 14 (14) | 11 (12)
BRONCHOPNEUMONIA (Infections and infestations) | 3 (3) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (3) | 3 (3)
PNEUMONIA (Infections and infestations) | 3 (3) | 2 (2)
INFECTED SKIN ULCER (Infections and infestations) | 2 (2) | 1 (1)
PURULENT DISCHARGE (Infections and infestations) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SHUNT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HYPOPHARYNGEAL CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 2 (2) | 2 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1)
DIABETIC COMA (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1)
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 11 (14) | 9 (9)
EXTREMITY NECROSIS (Vascular disorders) | 10 (11) | 9 (9)
NECROSIS ISCHAEMIC (Vascular disorders) | 6 (6) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 2 (2) | 0 (0)
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
ISCHAEMIA (Vascular disorders) | 1 (1) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprostadil (N=416) | Placebo (N=423)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 24 (29) | 26 (28)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 40 (41) | 41 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days